CLINICAL TRIAL: NCT07383285
Title: CAPOX and Bevacizumab With or Without Primary Tumor Radiotherapy and Iparomlimab and Tuvonralimab as First-line Treatment for RAS-Mutant/MSS Metastatic Rectal Cancer: An Open-label, Randomized, Multi-center Phase II Study
Brief Title: CAPOX and Bevacizumab With or Without Primary Tumor Radiotherapy and Iparomlimab and Tuvonralimab as First-line Treatment for RAS-Mutant/MSS Metastatic Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Shanxi Province Cancer Hospital (Other); West China Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Consultant, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOVA-Rec01
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rectal Neoplasms Malignant
MeSH Terms: interventions — Capecitabine; Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: Capox + Bev combined with primary lesion radiotherapy and (Iparomlimab and Tuvonralimab), administered once every 3 weeks (Q3w), for a maximum of 8 cycles. Then, it entered the maintenance treatment stage with Capecitabine + Bev + (Iparomlimab and Tuvonralimab), administered once every 3 weeks (Q3w).
  Interventions: Drug: Iparomlimab and Tuvonralimab; Radiation: Radiotherapy to the primary site; Drug: Capecitabine; Drug: Bevacizumab; Drug: Oxaliplatin injection
- Control group (Active Comparator): Control group: Capox + Bev, administered once every 3 weeks (Q3w), for a maximum of 8 cycles. Then, it entered the maintenance treatment stage with Capecitabine + Bev, administered once every 3 weeks (Q3w).
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Oxaliplatin injection

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — (Experimental group) PD-1/CTLA-4 Antibody
  Other Names: QL1706
  Arms: Experimental group
Radiation: Radiotherapy to the primary site — (Experimental group) Radiotherapy to the primary site of rectal
  Arms: Experimental group
Drug: Capecitabine — (both groups)
Drug: Bevacizumab — (both groups)
Drug: Oxaliplatin injection — (both groups)

SUMMARY:
Research objective: To compare the efficacy and safety of Capox + Bev versus Capox + Bev combined with primary site radiotherapy + (Iparomlimab and Tuvonralimab) as the first-line treatment for RAS Mutation/pMMR metastatic rectal cancer patients.

Study endpoint:

Primary endpoint: 12-month progression-free survival rate (PFSR)

Secondary endpoints:

* The objective response rate (ORR) and disease control rate (DCR) as determined by the investigator according to the RECIST 1.1 standard, time to response (TTR), duration of response (DOR), progression-free survival (PFS), 6-month progression-free survival rate (PFSR), overall survival (OS);
* The frequency and severity of adverse events (AEs) during treatment (NCI CTCAE 5.0).

This study will enroll 106 patients (stratification factors: presence or absence of liver metastasis; whether NED could be achieved). They were randomly assigned in a 1:1 ratio to:

The treatment group: Capox + Bev combined with primary site radiotherapy and (Iparomlimab and Tuvonralimab), administered every 3 weeks (Q3w), up to a maximum of 8 cycles, followed by a maintenance treatment stage of Capecitabine + Bev + (Iparomlimab and Tuvonralimab), administered every 3 weeks (Q3w).

The control group: Capox + Bev, administered every 3 weeks (Q3w), up to a maximum of 8 cycles, followed by a maintenance treatment stage of Capecitabine + Bev, administered every 3 weeks (Q3w).

DETAILED DESCRIPTION:
This study is an open-label, randomized controlled, multicenter phase II clinical trial, aiming to evaluate the efficacy and safety of the Capox + Bev combination (with or without concurrent primary lesion radiotherapy + (Iparomlimab and Tuvonralimab) as the first-line treatment for patients with RAS mutation/pMMR metastatic rectal cancer.

This study will enroll 106 patients, (stratification factors: presence or absence of liver metastasis; whether NED could be achieved) and was randomly assigned in a 1:1 ratio to:

The treatment group: Capox + Bev combined with primary lesion radiotherapy and (Iparomlimab and Tuvonralimab), administered once every 3 weeks (Q3w), for a maximum of 8 cycles, followed by a maintenance treatment stage of Capecitabine + Bev + (Iparomlimab and Tuvonralimab), administered once every 3 weeks (Q3w).

The control group: Capox + Bev, administered once every 3 weeks (Q3w), for a maximum of 8 cycles, followed by a maintenance treatment stage of Capecitabine + Bev, administered once every 3 weeks (Q3w).

Treatment plan The experimental group will receive Capox + Bev combined with primary lesion radiotherapy and (Iparomlimab and Tuvonralimab): Oxaliplatin 130mg/m2 on day 1, Capecitabine 1000mg/m2 twice daily from day 1 to day 14, Bevacizumab 7.5mg/kg on day 1, (Iparomlimab and Tuvonralimab) 5mg/kg on day 1, repeated every 3 weeks, up to a maximum of 8 cycles. On the third cycle, primary lesion radiotherapy is conducted simultaneously, with the specific range and dose of 95% PGTV (rectal primary lesion) 25Gy/5 fractions [Before and after radiotherapy, the chemotherapy and Bevacizumab can be adjusted (stopped or reduced) according to the specific patient's adverse reactions]. Then enter the Capecitabine + Bev + (Iparomlimab and Tuvonralimab) maintenance treatment: Capecitabine 1000mg/m2 twice daily from day 1 to day 14, Bevacizumab 7.5mg/kg on day 1, (Iparomlimab and Tuvonralimab) 5mg/kg on day 1, repeated every 3 weeks. Until disease progression, occurrence of intolerable toxicity, acceptance of new anti-tumor treatment, withdrawal of informed consent, loss to follow-up, death, or other researchers determine that treatment should be stopped, whichever occurs first. If during the treatment process, one drug is discontinued for any reason, other drugs can continue to be used.

The control group will receive Capox + Bev: Oxaliplatin 130mg/m2 on day 1, Capecitabine 1000mg/m2 twice daily from day 1 to day 14, Bevacizumab 7.5mg/kg on day 1, repeated every 3 weeks, up to a maximum of 8 cycles. Then enter the Capecitabine + Bev maintenance treatment: Capecitabine 1000mg/m2 twice daily from day 1 to day 14, Bevacizumab 7.5mg/kg on day 1, repeated every 3 weeks. Until disease progression, occurrence of intolerable toxicity, acceptance of new anti-tumor treatment, withdrawal of informed consent, loss to follow-up, death, or other researchers determine that treatment should be stopped, whichever occurs first. If during the treatment process, one drug is discontinued for any reason, other drugs can continue to be used.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were able to understand the informed consent form, voluntarily participated and signed the informed consent form;
2. On the day of signing the informed consent form, the subjects were aged between 18 and 75 years old, regardless of gender;
3. Pathological tissue diagnosis confirmed rectal adenocarcinoma (including signet ring cell carcinoma and mucinous adenocarcinoma);
4. The lower boundary of the lesion was within 15 cm from the anal verge;
5. The clinical stage was stage IV;
6. The genetic test results were KRAS or NRAS mutations, without BRAF V600 mutations, and the immunohistochemical results were pMMR;
7. The subjects had not received palliative drug treatment, or had received 1 cycle of FOLFOX/CAPOX and had not undergone tumor efficacy assessment;
8. According to the RECIST 1.1 standard, there was at least 1 measurable lesion or assessable lesion at the baseline;
9. The primary lesion existed and had not undergone radiotherapy previously;
10. The ECOG score was 0 or 1 (Appendix 4);
11. The expected survival period was ≥ 6 months;
12. Female subjects with fertility or male subjects whose partner had fertility agreed to adopt effective contraceptive measures starting from 7 days before the first administration until 120 days after the last administration (refer to Appendix 3);
13. The subjects were capable and willing to comply with the visit, treatment plan, laboratory tests and other research-related procedures stipulated in the research protocol;
14. Within 7 days before the first administration, they had good organ function

Exclusion Criteria:

(1) Subjects with untreated active brain metastases or meningeal metastases; if the brain metastases of the subject have been treated and the condition of the metastases is stable (brain imaging examination at least 4 weeks before the first administration shows stable lesions, and there are no new neurological symptoms or the neurological symptoms have recovered to baseline levels), and there is no evidence of new onset or enlargement of the metastases, they are allowed to be enrolled; (2) Have the following cardiovascular conditions:

1. Active coronary heart disease with angina pectoris or patients who need to take medication to prevent angina attacks;
2. NYHA II-IV grade chronic heart failure;
3. Uncontrolled hypertension after drug treatment (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
4. Major vascular diseases (such as aortic aneurysm, aortic dissection aneurysm, internal carotid artery stenosis);
5. Has had thromboembolic or cerebrovascular embolic events within 6 months. (3) Have the following digestive system diseases:

1) Within 6 months, there has been abdominal fistula, gastrointestinal perforation or abdominal abscess or active gastrointestinal bleeding. If the perforation or fistula has been treated by resection or repair, and the disease has been judged by the investigator to have recovered or alleviated, it is allowed to be enrolled; 2) Have gastric, duodenal ulcers or ulcer malignancy, intestinal obstruction/obstruction with incomplete obstruction; 3) Have chronic enteritis and/or inflammatory bowel disease; (4) Have abnormal coagulation conditions:

1. Have bleeding (including hemoptysis) or coagulation disorders;
2. Are taking warfarin, aspirin (except for small doses of less than 100 mg per day), low molecular weight heparin and other antiplatelet aggregation Chinese and Western drugs.

(5) Within 28 days before the first administration or 5 half-lives (whichever is shorter, but at least 2 weeks) have received any other interventional clinical trials or received other anti-tumor treatment for the purpose of alleviating symptoms of bone metastases is allowed; (6) Within 28 days before the first administration have received major surgical treatment (such as major surgeries through the abdomen or thorax; excluding drainage, diagnostic punctures or peripheral vascular access replacement surgeries); (7) Within 14 days before the first administration need to receive continuous 7 days of systemic corticosteroid treatment (≥ 10 mg/day prednisone, or equivalent other corticosteroids) or immunosuppressant treatment; except for inhalation or local application of corticosteroids, or receiving physiological replacement doses of corticosteroids due to adrenal insufficiency; allowed for short-term (≤ 7 days) corticosteroids for prevention (for example, contrast agent allergy) or treatment of non-autoimmune diseases (for example, delayed-type hypersensitivity reaction caused by exposure to allergens); (8) Within 28 days before the first administration have received live vaccines (including attenuated live vaccines); (9) Have interstitial lung disease, or have a history of non-infectious pneumonia requiring oral or intravenous administration of glucocorticoids; (10) Within 2 years before the start of the study treatment need systemic treatment for active autoimmune diseases, or the investigator judges that there is a possibility of recurrence or planned treatment for autoimmune diseases. The following are excluded: a) Skin diseases that do not require systemic treatment (such as: vitiligo, alopecia, psoriasis or eczema); b) Hypothyroidism caused by autoimmune thyroiditis, only requiring stable doses of hormone replacement therapy; c) Type I diabetes that only requires stable doses of insulin replacement therapy; d) Childhood asthma has completely resolved, and no intervention is needed after adulthood; e) The investigator judges that the disease will not recur without external triggering factors. (11) Within 5 years prior to the first administration, having another malignant tumor, except for cured skin squamous cell carcinoma, basal cell carcinoma, non-invasive bladder cancer, localized low-risk prostate cancer (defined as stage ≤ T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL at the time of prostate cancer diagnosis (if measured), patients who have received radical treatment and have no biochemical recurrence of prostate-specific antigen (PSA)), and in situ cervical/breast cancer; (12) Having uncontrolled comorbidities, including but not limited to the following conditions: a) Active HBV or HCV infection; b) Subjects with positive HBsAg and/or HCV antibody during the screening period, must undergo HBV DNA and/or HCV RNA testing. Subjects with HBV DNA ≤ 500 IU/mL (or ≤ 2000 copies/mL) and/or negative HCV RNA can be enrolled; during the trial, the study investigator decides to monitor HBV DNA based on the subject's condition; c) Known HIV infection or AIDS history; d) Active tuberculosis; e) Active infection or systemic use of anti-infective drugs for more than 1 week before the first administration of this study and within 28 days before the first administration; fever of unknown origin occurred within 2 weeks before administration; f) Uncontrolled hypertension (resting blood pressure ≥ 160/100 mmHg), symptomatic heart dysfunction (NYHA II-IV), unstable angina pectoris or myocardial infarction within 6 months, or QTc prolongation or risk of arrhythmia (baseline QTc > 470 msec corrected by Fridericia method, refractory hypokalemia, long QT syndrome, resting heart rate > 100 bpm atrial fibrillation or severe valvular heart disease); g) Active bleeding that cannot be controlled by medical treatment; (13) Toxicity from previous anti-tumor therapy has not recovered to CTCAE ≤ 1 grade (NCI-CTCAE v5.0) or baseline level, except alopecia, skin pigmentation (allowing any grade), and immune-related adverse reactions that require physiological dose substitution (such as hypothyroidism, pituitary insufficiency, type I diabetes, etc.); (14) Previous history of allogeneic bone marrow or organ transplantation; (15) Previous history of allergic reactions to antibody drugs, hypersensitivity reactions, or intolerance (such as severe allergic reactions, immune-mediated liver toxicity, immune-mediated thrombocytopenia or anemia); (16) Pregnant and/or lactating women; (17) Other situations that the investigator considers to affect the safety or compliance of the treatment with the study drug, including but not limited to moderate to large pleural/abdominal effusion/pericardial effusion, refractory pleural/abdominal effusion/pericardial effusion, intestinal obstruction or subacute intestinal obstruction, mental disorders, etc.; (18) Previous treatment with immune checkpoint blockers or T-cell co-stimulation drugs, including but not limited to immune checkpoint blockers such as PD-1, PD-L1, CTLA4, LAG3, etc., therapeutic vaccines, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
12-month disease-free survival rate (progression-free survival rate, PFSR) | From randomization to disease progression or death from any cause, whichever occurs first; the progression-free survival rate will be estimated at 12 months.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From randomization to the first documented tumor response, assessed during the entire treatment period and follow-up, up to 24 months.
Disease control rate (DCR) | From randomization to the first documented tumor response, assessed during the entire treatment period and follow-up, up to 24 months.
Time to response (TTR) | From randomization to the first documented objective response (complete or partial response), assessed up to 24 months.
Duration of response (DOR) | From the first documented objective response (CR or PR) to disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
6-month progression-free survival rate (PFSR) | From randomization to disease progression or death from any cause, whichever occurs first; the progression-free survival rate will be estimated at 6 months.
Progression-free survival (PFS) | From randomization to disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
Overall survival (OS) | From randomization to death from any cause, assessed up to 24 months.